CLINICAL TRIAL: NCT02090348
Title: A Multicenter, Open-Label Study to Evaluate Fatigue in Subjects With Relapsing-Remitting Multiple Sclerosis During Treatment With Tecfidera® (Dimethyl Fumarate) Gastro-Resistant Hard Capsules (TECNERGY)
Brief Title: Study to Evaluate Fatigue in Participants With Relapsing Remitting Multiple Sclerosis When Treated With Dimethyl Fumarate
Acronym: TECNERGY
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was withdrawn for business reasons. The decision to stop the TECNERGY study was not a result of any safety or efficacy concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109MS405; 2013-001025-53 (EudraCT Number); DEN-BGT-13-10413 (Other: Biogen)
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dimethyl fumarate (Experimental): DMF at a dose of 120 mg twice a day (BID) for the first 7 days and 240 mg BID for the remainder of study period (up to 12 months)
  Interventions: Drug: dimethyl fumarate

INTERVENTIONS:
Drug: dimethyl fumarate — Administered as specified in the treatment arm
  Other Names: DMF; BG00012; Tecfidera

SUMMARY:
The primary objective of this study is to determine whether dimethyl fumarate (DMF) taken over 12 months is effective in reducing Multiple Sclerosis (MS)-related fatigue, as measured by mean changes in the Fatigue Scale for Motor and Cognitive Functions (FSMC), in participants with relapsing-remitting multiple sclerosis (RRMS). The secondary objectives of this study are: To investigate changes from Baseline in FSMC and fatigue severity (Fatigue Severity Scale [FSS]) at 1, 3, 6, 9, and 12 months in participants receiving DMF; To assess the impact of DMF on patient-reported outcomes (PROs), including work productivity (Work Productivity and Activity Impairment-Multiple Sclerosis questionnaire [WPAI-MS]), health-related quality of life (Short Form Health Survey [SF-12]), depression (Beck Depression Inventory-Fast Screen [BDI-FS]), and sleepiness (Epworth Sleepiness Scale [ESS]) at 6 and 12 months in participants receiving DMF; To examine whether an association exists between fatigue and baseline demographics (e.g., age and sex) and disease characteristics (e.g., disease duration, baseline disease activity, treatment history, expanded disability status scale [EDSS] score, and PROs); To assess any changes in fatigue-related medication use.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a confirmed diagnosis of RRMS and satisfies the therapeutic indication as described in the local label.
* Have a stable EDSS (as assessed by the Investigator) and been on the same (type and dosage) standard of care (SOC) first-line treatment for at least 6 months.
* If taking antidepressants, amphetamine, modafinil, or fampridine (Fampyra), subject must be assessed as having been clinically stable for at least 3 months prior to the Baseline Visit.
* FSMC total score ≥43 (mild fatigue) at Baseline.
* As perceived by the Investigator, have the ability to comply with all requirements of the study protocol.

Key Exclusion Criteria:

* Diagnosis of major depression, as identified by the Investigator.
* Diagnosis of primary progressive, secondary progressive, or progressive relapsing multiple sclerosis.
* History of malignancy (except for basal cell carcinoma that had been completely excised prior to study entry), severe allergic or anaphylactic reactions or known drug hypersensitivity, abnormal laboratory results indicative of any significant disease, and/or a major disease that would preclude participation in a clinical trial.
* Treatment of MS relapse within 90 days prior to study enrollment.
* History of a positive test result for human immunodeficiency virus, hepatitis C virus antibody, or hepatitis B virus (defined as positive for hepatitis B surface antigen or hepatitis B core antibody.
* Impaired hepatic or renal function, as perceived by the Investigator.
* Any prior treatment with DMF (or other fumarate derivative), total lymphoid irradiation, cladribine, fingolimod, T cell or T-cell receptor vaccination, or any therapeutic monoclonal antibody.
* Current enrollment in any other clinical studies.
* Known to suffer from narcolepsy or another significant sleep disorder.
* Comorbidity that may have an impact on fatigue.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen Idec, make the subject unsuitable for enrollment.

NOTE: Other protocol-defined Inclusion/Exclusion Criteria May Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in MS-related fatigue as assessed by FSMC at 12 months in participants receiving DMF | 12 months
  FSMC is a 20-item questionnaire and produces a score between 1 and 5 for each scored question (ranging from "does not apply at all" to "applies completely"). Items are summed to generate a total score and transformed to a scale with a range of 20 to 100, where higher scores indicate higher levels of fatigue

SECONDARY OUTCOMES:
Mean change from baseline in fatigue as assessed by FSMC in participants receiving DMF | Baseline and 1, 3, 6, 9 and 12 months
Mean change from baseline in fatigue as assessed by FSS in participants receiving DMF | Baseline and 1, 3, 6, 9 and 12 months
  The Fatigue Severity Scale (FSS) is designed to differentiate fatigue from clinical depression, since both share some of the same symptoms. FSS consists of answering a 9-item questionnaire that requires the participant to rate his or her own level of fatigue. Each question produces a score between 1 to 7. The scoring is done by calculating the average response to the questions. Participants with depression alone score about 4.5. But people with fatigue related to MS average about 6.5
Mean change from baseline in work productivity as assessed by WPAI-MS, in participants receiving DMF | Baseline and 6, 12 months
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity
Mean change from baseline in quality of life as assessed by SF-12 in participants receiving DMF | Baseline and 6, 12 months
  The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health
Mean change from baseline in depression as assessed by BDI-FS in participants receiving DMF | Baseline and 6, 12 months
  BDI-FS is a self-report inventory for measuring the severity of depression on a 7-item questionnaire. Each question is rated on a 4-point scale (0 - 3) to assess frequency, over the past two weeks, of feelings of sadness, pessimism (hopelessness), sense of failure, loss of a sense of pleasure, loss of self-confidence, self-blame, and suicidal ideation. The total ESS score is the sum of 8 item-scores and can range between 0 and 21, where higher scores indicate higher levels of depression
Mean change from baseline in sleepiness assessed by ESS in participants receiving DMF | Baseline and 6, 12 months
  The ESS is a self-administered 8-item questionnaire with that provides a measure of a person's general level of daytime sleepiness, or their average sleep propensity in daily life. Each question is rated on a 4-point scale (0 - 3), their usual chances of dozing off or falling asleep in 8 different situations or activities that most people engage in as part of their daily lives, although not necessarily every day. The total ESS score is the sum of 8 item-scores and can range between 0 and 24, where higher scores indicate higher levels of a person's level of daytime sleepiness
Change in MS-related fatigue (FSMC) status | Baseline and up to 12 months
  Improved (> 4.5 increase), Stable (within ±4.5), and Worsened (> 4.5 decrease)
Correlation of fatigue with baseline demographics and disease characteristics | Baseline and up to 12 months
Proportion of participants with reduced dose or discontinuation of fatigue-related medications | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen